CLINICAL TRIAL: NCT07266428
Title: Phase 1/2A Study of OTP-01, a Dual Paratopic PD-1/VEGFR2 Antibody, in Patients With Advanced Solid Tumors
Brief Title: A Study of OTP-01, a Dual Paratopic PD-1/VEGFR2 Antibody, in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ottimo Pharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: OTP-01-101; 2025-524111-37-00 (EU CTIS Number); U1111-1329-6711 (Other: WHO)
Record Dates: First submitted 2025-11-16; First posted 2025-12-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
Keywords: advanced solid tumors

STUDY DESIGN:
Intervention Model Description: Phase 1 monotherapy dose escalation with backfill followed by Phase 2A monotherapy dose expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Monotherapy Dose Escalation with Backfill (Experimental)
  Interventions: Drug: OTP-01
- Monotherapy Dose Expansion (Experimental)
  Interventions: Drug: OTP-01

INTERVENTIONS:
Drug: OTP-01 — Intravenous (IV) Infusion

SUMMARY:
The main goals of this clinical trial are to find out what the best dose of the study drug, OTP-01, is for patients with solid tumors through understanding how it is tolerated and any side effects that it may cause. The trial will also see if OTP-01 causes tumors to shrink and how the body processes OTP-01 by measuring drug levels in the blood.

The main questions this study aims to answer are:

* What is the recommended dose of OTP-01 for adults with solid tumors?
* Is OTP-01 safe and tolerable?
* Does OTP-01 reduce tumor growth?

Participants will:

* Receive OTP-01 through an infusion into a vein. Doses will be spaced out and never more than once a week.
* Have blood tests to evaluate safety and drug levels of OTP-01. These will be done often at first and then less frequently as treatment continues.
* Have radiographic scans of their tumor at baseline and during the study at regular intervals.
* Have the choice to have an optional tumor biopsy before and after treatment to help researchers understand how OTP-01 affects cancer and the immune system. These biopsies are voluntary and will not affect participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced (incurable, recurrent, unresectable, or metastatic) solid tumors.

   1. For dose escalation cohort patients: patients must have a tumor type as defined in the protocol. Patients will have progression on or after or intolerance to most recent systemic therapy. Patients must have received approved standard therapy that is available to the patient that is known to confer clinical benefit, unless this therapy is contraindicated, intolerable to the patient, or is declined by the patient. The reason for treatment decline must be clearly documented in the medical record.
   2. For backfill cohorts: patients must have a tumor type as defined in the protocol. If patients decline an available standard therapeutic regimen known to confer benefit to enroll on this study, the discussion must be clearly documented in the medical record.
2. Measurable disease per RECIST v1.1. Additionally, patients with breast or ovarian cancer with non-measurable, evaluable disease are eligible.
3. ECOG performance status 0-1.
4. Life expectancy of at least 3 months.
5. Willing to provide a pretreatment tumor sample (either an archival sample or a sample obtained by pretreatment biopsy).
6. All toxicity resulting from prior cancer therapies must have resolved to NCI CTCAE v5.0 ≤ Grade 1 or pre-therapy baseline with the exception of alopecia or ≤ Grade 2 neuropathy.
7. Adequate hematological, renal, and hepatic function.
8. Other protocol-defined inclusion criteria apply.

Exclusion Criteria:

1. Receiving systemic corticosteroids at prednisone-equivalent dose of > 10 mg/day within 4 weeks prior to signing consent. Chronic systemic corticosteroid therapy for physiologic replacement (≤ 10 mg/day of prednisone equivalents) and the use of non-systemic corticosteroids (e.g., inhaled, topical, intra-nasal, intra-articular, or ophthalmic) are permitted
2. History of Grade 4 allergic or anaphylactic reaction to prior monoclonal antibody therapy or allergic reaction to any excipients within the investigational product
3. History of toxicity requiring permanent discontinuation of prior cancer immunotherapy
4. Have an active autoimmune disease that has required systemic treatment in past 2 years (replacement therapy is not considered a form of systemic treatment)
5. History of organ or stem cell transplant or need for immunosuppressive treatment
6. Have proteinuria > 2 + (within 7 days prior to initiation of study treatment).
7. Received any chemotherapy, immunotherapy or investigational anticancer therapy within 3 weeks or 5 half-lives (whichever is shorter; minimum of 2 weeks) prior to first dose of study drug
8. Definitive radiotherapy within 6 weeks and palliative radiation within 2 weeks prior to the first dose of study drug. If previously irradiated, lesions must have demonstrated clear-cut progression prior to being eligible for evaluation as target lesions
9. Other protocol and subprotocol-defined exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1 and Phase 2A: Frequency and Severity of adverse events (AEs) and serious adverse events (SAEs) | C1D1 through EoT (up to 36 months)
Phase 2A - Progression Free Survival (PFS) | C1D1 through EoT (up to 36 months)
Phase 2A - Disease Control Rate (DCR) | C1D1 through EoT (up to 36 months)
Phase 2A - Duration of Response (DOR) | C1D1 through EoT (up to 36 months)
Phase 2A - Objective Response Rate (ORR) | C1D1 through EoT (up to 36 months)

SECONDARY OUTCOMES:
Phase 1 and Phase 2A - plasma concentrations of OTP-01 | C1D1 through EOT (up to 36 months)
  As a function of time post-dosing
Phase 1 and Phase 2A - Area under the curve [AUC] | C1D1 through EOT (up to 36 months)
Phase 1 and Phase 2A - Maximum plasma concentration [Cmax] | C1D1 through EOT (up to 36 months)
Phase 1 and Phase 2A - Minimum plasma concentration [Cmin] | C1D1 through EOT (up to 36 months)
Phase 1 and Phase 2A - Time of maximum concentration [Tmax] | C1D1 through EOT (up to 36 months)
Phase 1 and Phase 2A - Half-life [t1/2] | C1D1 through EOT (up to 36 months)
Phase 1 and Phase 2A - Clearance [CL] | C1D1 through EOT (up to 36 months)
Phase 1 - Progression Free Survival (PFS) | C1D1 through EoT (up to 36 months)
Phase 1 - Disease Control Rate (DCR) | C1D1 through EoT (up to 36 months)
Phase 1 - Duration of Response (DOR) | C1D1 through EoT (up to 36 months)
Phase 1 - Objective Response Rate (ORR) | C1D1 through EoT (up to 36 months)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bell-McGuinn, Study Director — Ottimo Pharma Limited
Locations (4):
- United States (3):
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
- Linear Clinical Research, Nedlands, Australia

IPD SHARING:
Plan to Share IPD: Undecided